CLINICAL TRIAL: NCT07136909
Title: Validation of the French Version of the OSA-18 Questionnaire
Acronym: French OSA18
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0721
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Apnea, Obstructive
Keywords: Obstructive sleep apnea; sleep disordered breathing; questionnaire
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children referred to the sleep clinic for polysomnography.: Children aged 4 to 17 years referred hospitalized in the sleep unit of the Hospices Civils de Lyon (France) for polysomnography, for a duration of 24 to 48h.
  Interventions: Other: Completion of the OSA-18 questionnaire by parents, during hospitalization planned as part of routine care.

INTERVENTIONS:
Other: Completion of the OSA-18 questionnaire by parents, during hospitalization planned as part of routine care. — Completion of the OSA-18 questionnaire by parents, during hospitalization planned as part of routine care.

SUMMARY:
Obstructive sleep apnea (OSA) is characterized by repetitive partial and/or total closure of the upper airway during sleep, inducing oxygen desaturation and sleep disturbance. Its prevalence in the pediatric population is 1-5%. In children, OSA can have negative consequences on the cardiovascular system and on the neurocognitive development. It is essential to diagnose OSA and to treat it efficiently.

The OSA-18 questionnaire assesses the symptômes of OSA in children and its repercussions. It is composed of 18 items scored on a Likert scale by caregivers. This system allows a more sensitive scoring than binary answers available in other questionnaires like the Pediatric Sleep Questionnaire.

The OSA-18 questionnaire would thus be an interesting tool to use for evaluating treatment efficacy in interventional studies and in clinical practice.

This questionnaire is not yet available in French. The main objective of this study is thus to evaluate the validity of a French version compared to the gold standard method to evaluate OSA: polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized in the Clinical Epileptology, Sleep Disorders, and Child Functional Neurology Department for polysomnography to screen for OSA,
* Aged 4 to 17 years inclusive.

Exclusion Criteria:

* Parents and/or children object to participation in the study.
* Subjects participating in another intervention research study with an ongoing exclusion period.

Ages: 4 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Children aged 4 to 17 years referred hospitalized in the sleep unit of the Hospices Civils de Lyon (France) for polysomnography, for a duration of 24 to 48h.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Scores on the French version of the OSA-18 questionnaire (total score) | Day 2
  The OSA-18 questionnaire will be filled-in by caregivers.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme-Mère-Enfant, Bron, Rhône, France

IPD SHARING:
Plan to Share IPD: No